CLINICAL TRIAL: NCT03766581
Title: A Global, Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study of BMS-986177, an Oral Factor XIa Inhibitor, for the Prevention of New Ischemic Stroke or New Covert Brain Infarction in Patients Receiving Aspirin and Clopidogrel Following Acute Ischemic Stroke or Transient Ischemic Attack (TIA)
Brief Title: A Study on BMS-986177 for the Prevention of a Stroke in Patients Receiving Aspirin and Clopidogrel
Acronym: AXIOMATIC-SSP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CV010-031
Record Dates: First submitted 2018-11-13; First posted 2018-12-06 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Acute Ischemic Stroke; Transient Ischemic Attack (TIA)
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient | interventions — milvexian; Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- BMS-986177 Placebo (Placebo Comparator): Specified Dose on Specified Days
  Interventions: Other: Placebo; Drug: Clopidogrel; Drug: Aspirin
- Dose 1: BMS-986177 + Aspirin + Clopidogrel (Experimental): Specified Dose on Specified Days
  Interventions: Drug: BMS-986177; Drug: Clopidogrel; Drug: Aspirin
- Dose 2: BMS-986177 + Aspirin + Clopidogrel (Experimental): Specified Dose on Specified Days
  Interventions: Drug: BMS-986177; Drug: Clopidogrel; Drug: Aspirin
- Dose 3: BMS-986177 + Aspirin + Clopidogrel (Experimental): Specified Dose on Specified Days
  Interventions: Drug: BMS-986177; Drug: Clopidogrel; Drug: Aspirin
- Dose 4: BMS-986177 + Aspirin + Clopidogrel (Experimental): Specified Dose on Specified Days
  Interventions: Drug: BMS-986177; Drug: Clopidogrel; Drug: Aspirin
- Dose 5: BMS-986177 + Aspirin + Clopidogrel (Experimental): Specified Dose on Specified Days
  Interventions: Drug: BMS-986177; Drug: Clopidogrel; Drug: Aspirin
- Dose 6: BMS-986177 + Aspirin + Clopidogrel (Experimental): Specified Dose on Specified Days
  Interventions: Drug: BMS-986177; Drug: Clopidogrel; Drug: Aspirin
- Dose 7: BMS-986177 + Aspirin + Clopidogrel (Experimental): Specified Dose on Specified Days
  Interventions: Drug: BMS-986177; Drug: Clopidogrel; Drug: Aspirin

INTERVENTIONS:
Drug: BMS-986177 — Oral administration
  Arms: Dose 1: BMS-986177 + Aspirin + Clopidogrel; Dose 2: BMS-986177 + Aspirin + Clopidogrel; Dose 3: BMS-986177 + Aspirin + Clopidogrel; Dose 4: BMS-986177 + Aspirin + Clopidogrel; Dose 5: BMS-986177 + Aspirin + Clopidogrel; Dose 6: BMS-986177 + Aspirin + Clopidogrel; Dose 7: BMS-986177 + Aspirin + Clopidogrel
Other: Placebo — Oral Administration
  Arms: BMS-986177 Placebo
Drug: Clopidogrel — Oral administration
Drug: Aspirin — Oral administration

SUMMARY:
The purpose of this clinical study is to determine whether the addition of an oral Factor XIa Inhibitor to Aspirin and Clopidogrel is more effective than standard therapy in secondary stroke prevention.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female ≥40 years of age
* Acute Ischemic Stroke or Transient Ischemic Attack
* Intracranial or Extracranial Atherosclerotic Plaque proximal to the affected brain area

Exclusion Criteria:

* Predicted inability to swallow study medication
* Any condition that, in the opinion of the Investigator, contraindicates anticoagulant therapy or would have an unacceptable risk of bleeding
* Use of thrombolytic therapy or mechanical thrombectomy for treatment of index stroke

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2366 (Actual)
Dates: Start 2019-01-27 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (421):
- United States (65):
  - Local Institution - 0029, Birmingham, Alabama
  - Local Institution - 0007, Glendale, California
  - Local Institution - 0006, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Local Institution - 0231, Los Angeles, California
  - Local Institution - 0376, Sacramento, California
  - Local Institution - 0004, Stanford, California
  - Local Institution - 0042, Torrance, California
  - Local Institution - 0340, Newark, Delaware
  - Local Institution - 0075, Gainesville, Florida
  - Local Institution - 0013, Sarasota, Florida
  - Local Institution - 0024, Tampa, Florida
  - Local Institution - 0015, Augusta, Georgia
  - Local Institution - 0428, Honolulu, Hawaii
  - Local Institution - 0293, Chicago, Illinois
  - University of Illinois Hospital & Health Sciences System, Chicago, Illinois
  - Local Institution - 0430, Elk Grove Village, Illinois
  - Local Institution - 0382, Rockford, Illinois
  - Local Institution - 0346, Louisville, Kentucky
  - Local Institution - 0047, New Orleans, Louisiana
  - Local Institution - 0420, Baltimore, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution - 0236, Boston, Massachusetts
  - Local Institution, Detroit, Michigan
  - Local Institution - 0434, Detroit, Michigan
  - Local Institution - 0375, Farmington Hills, Michigan
  - Local Institution, Minneapolis, Minnesota
  - Local Institution, Kansas City, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution - 0294, St Louis, Missouri
  - Local Institution - 0352, St Louis, Missouri
  - Advanced Neurology Specialists PLLC, Great Falls, Montana
  - Local Institution - 0276, Camden, New Jersey
  - Local Institution - 0039, New Brunswick, New Jersey
  - Local Institution - 0354, Brooklyn, New York
  - Local Institution, Buffalo, New York
  - Local Institution, New York, New York
  - Local Institution - 0125, New York, New York
  - Duke University Medical Center, Butner, North Carolina
  - Local Institution - 0043, Chapel Hill, North Carolina
  - Local Institution - 0016, Greensboro, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution - 0003, Cleveland, Ohio
  - Local Institution - 0050, Cleveland, Ohio
  - Local Institution - 0419, Columbus, Ohio
  - Local Institution - 0218, Oklahoma City, Oklahoma
  - Local Institution - 0022, Portland, Oregon
  - Local Institution - 0302, Abington, Pennsylvania
  - Local Institution, Allentown, Pennsylvania
  - Local Institution, Camp Hill, Pennsylvania
  - Local Institution - 0018, Erie, Pennsylvania
  - Local Institution - 0020, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Local Institution - 0019, York, Pennsylvania
  - Local Institution - 0041, Columbia, South Carolina
  - Local Institution - 0009, Nashville, Tennessee
  - Local Institution - 0008, Austin, Texas
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - Local Institution, Dallas, Texas
  - University Medical center of El Paso, El Paso, Texas
  - Local Institution - 0040, Houston, Texas
  - Local Institution - 0093, Houston, Texas
  - Local Institution - 0187, Temple, Texas
  - Local Institution, Richmond, Virginia
  - Local Institution, Milwaukee, Wisconsin
- Argentina (9):
  - Local Institution - 0100, Adrogué, Buenos Aires
  - Local Institution - 0063, CABA, Buenos Aires
  - Local Institution - 0076, CABA, Buenos Aires
  - Local Institution - 0067, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 0237, Lomas de Zamora, Buenos Aires
  - Local Institution - 0435, Recoleta, Buenos Aires
  - Local Institution, Buenos Aires
  - Local Institution - 0068, Buenos Aires
  - Local Institution, Santa Fe
- Australia (8):
  - Local Institution - 0329, Randwick, New South Wales
  - Local Institution - 0360, Sydney, New South Wales
  - Local Institution - 0287, Southport, Queensland
  - Local Institution - 0399, Adelaide, South Australia
  - Local Institution - 0397, Launceston, Tasmania
  - Local Institution - 0358, Clayton, Victoria
  - Local Institution - 0281, Heidelberg, Victoria
  - Local Institution - 0315, Murdoch, Western Australia
- Austria (4):
  - Local Institution - 0184, Klagenfurt
  - Local Institution, Sankt Pölten
  - Local Institution - 0273, Vienna
  - Local Institution - 0106, Vöcklabruck
- Belgium (12):
  - Local Institution - 0122, Edegem, Antwerpen
  - Local Institution - 0196, Brussels, Brussels Capital
  - Local Institution - 0192, Yvoir, Namur
  - Local Institution, Brasschaat
  - Local Institution - 0284, Bruges
  - Local Institution - 0427, Brussels
  - Local Institution - 0305, Brussels
  - Local Institution - 0190, Brussels
  - Local Institution - 0199, Ghent
  - Local Institution - 0103, Kortrijk
  - Local Institution - 0098, Leuven
  - Local Institution - 0178, Liège
- Brazil (11):
  - Local Institution - 0072, Fortaleza, Ceará
  - Local Institution - 0275, Uberaba, Minas Gerais
  - Local Institution - 0314, Curitiba, Paraná
  - Local Institution - 0200, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0219, Joinville, Santa Catarina
  - Local Institution - 0245, Botucatu, São Paulo
  - Local Institution - 0065, Campinas, São Paulo
  - Local Institution, Ribeirão Preto, São Paulo
  - Local Institution - 0113, Santo André, São Paulo
  - Local Institution - 0234, São Paulo, São Paulo
  - Local Institution - 0248, São Paulo, São Paulo
- Canada (14):
  - Local Institution - 0057, Calgary, Alberta
  - Local Institution - 0061, Edmonton, Alberta
  - Local Institution - 0059, Lethbridge, Alberta
  - Local Institution - 0369, New Westminster, British Columbia
  - Local Institution - 0121, Vancouver, British Columbia
  - Local Institution - 0054, Hamilton, Ontario
  - Local Institution, Kingston, Ontario
  - Local Institution - 0227, London, Ontario
  - Local Institution - 0124, Toronto, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution - 0326, Chicoutimi, Quebec
  - Local Institution - 0155, Greenfield Park, Quebec
  - Local Institution - 0066, Montreal, Quebec
  - Local Institution - 0064, Québec, Quebec
- Chile (4):
  - Local Institution - 0172, Viña del Mar, Región de Valparaíso
  - Local Institution, Los Ángeles
  - Local Institution - 0131, Valdivia
  - Local Institution - 0167, Viña del Mar
- China (12):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Haikou, Hainan
  - Local Institution, Daqing, Heilongjiang
  - Local Institution, Zhengzhou, Henan
  - Local Institution, Nantong, Jiangsu
  - Local Institution, Yangzhou, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Shenyang, Liaoning
  - Local Institution, Qingdao, Shandong
  - Local Institution, Yantai, Shandong
  - Local Institution, Wenzhou, Zhejiang
- Czechia (6):
  - Local Institution - 0348, Jihlava, Kraj Vysočina
  - Local Institution - 0401, Olomouc, Olomoucký kraj
  - Local Institution, Brno
  - Local Institution, České Budějovice
  - Local Institution - 0023, Ostrava
  - Local Institution - 0339, Prague
- Denmark (5):
  - Local Institution - 0117, Herlev, Capital
  - Local Institution - 0217, Aalborg
  - Local Institution - 0127, Aarhus N
  - Local Institution - 0142, Copenhagen
  - Local Institution - 0110, Glostrup Municipality
- Finland (3):
  - Local Institution - 0111, Helsinki
  - Local Institution - 0341, Lappeenranta
  - Local Institution - 0143, Turku
- France (17):
  - Local Institution - 0442, Montpellier, Hérault
  - Local Institution - 0048, Lille, Nord
  - Local Institution - 0051, Bordeaux
  - Local Institution, Bourg-en-Bresse
  - Local Institution - 0165, Brest
  - Local Institution - 0174, Caen
  - Local Institution, Créteil
  - Local Institution, Limoges
  - Local Institution - 0168, Marseille
  - Local Institution - 0297, Nancy
  - Local Institution - 0205, Nîmes
  - Local Institution - 0049, Paris
  - Local Institution, Paris
  - Local Institution - 0126, Paris
  - Local Institution - 0028, Paris
  - Local Institution - 0107, Rouen
  - Local Institution - 0355, Toulouse
- Germany (29):
  - Local Institution - 0391, Sindelfingen, Baden-Wurttemberg
  - Local Institution - 0045, Tübingen, Baden-Wurttemberg
  - Local Institution - 0285, Frankfurt am Main, Hesse
  - Local Institution - 0090, Leipzig, Saxony
  - Local Institution - 0258, Lübeck, Schleswig-Holstein
  - Local Institution - 0011, Altenburg
  - Local Institution - 0032, Berlin
  - Local Institution, Berlin
  - Local Institution, Bielefeld
  - Local Institution - 0250, Bonn
  - Local Institution - 0380, Bremen
  - Local Institution - 0144, Dresden
  - Local Institution - 0097, Erlangen
  - Local Institution - 0053, Essen
  - Local Institution - 0291, Frankfurt am Main
  - Local Institution - 0254, Giessen
  - Local Institution - 0056, Hamburg
  - Local Institution - 0044, Hamburg
  - Local Institution - 0034, Hamburg
  - Local Institution, Hanover
  - Local Institution - 0055, Heidelberg
  - Local Institution, Magdeburg
  - Local Institution - 0036, Minden
  - Local Institution - 0256, Münster
  - Local Institution - 0378, Osnabrück
  - Local Institution - 0367, Regensburg
  - Local Institution - 0387, Sande
  - Local Institution, Siegen
  - Local Institution - 0241, Ulm
- Greece (25):
  - Local Institution - 0438, Athens, Attica
  - Local Institution - 0357, Larissa, Larisa
  - Local Institution - 0370, Athens
  - Local Institution - 0436, Athens
  - Local Institution - 0440, Athens
  - Local Institution - 0373, Athens
  - Local Institution, Athens
  - Local Institution - 0209, Athens
  - Local Institution - 0283, Athens
  - Local Institution - 0351, Athens
  - Local Institution - 0407, Crete
  - Local Institution, Ioannina
  - Local Institution - 0161, Larissa
  - Local Institution - 0441, Larissa
  - Local Institution - 0333, Loanniana
  - Local Institution - 0365, Loanniana
  - Local Institution - 0439, Neo Faliro
  - Local Institution - 0371, Pátrai
  - Local Institution - 0208, Pireaus
  - Local Institution - 0405, Thessaloniki
  - Local Institution - 0269, Thessaloniki
  - Local Institution - 0389, Thessaloniki
  - Local Institution - 0444, Thessaloniki
  - Local Institution - 0210, Thessaloniki
  - Local Institution - 0445, Thessaloniki
- Local Institution, Hong Kong, Hong Kong
- Hungary (13):
  - Local Institution - 0070, Miskolc, BZ
  - Local Institution - 0134, Budapest
  - Local Institution - 0077, Budapest
  - Local Institution - 0119, Budapest
  - Local Institution - 0136, Budapest
  - Local Institution - 0154, Debrecen
  - Local Institution - 0079, Győr
  - Local Institution - 0175, Kistarcsa
  - Local Institution - 0437, Kisvárda
  - Local Institution - 0220, Nyíregyháza
  - Local Institution - 0138, Pécs
  - Local Institution - 0133, Szeged
  - Local Institution - 0137, Zalaegerszeg
- Israel (10):
  - Local Institution, Beersheba
  - Local Institution - 0139, Haifa
  - Local Institution - 0349, Haifa
  - Local Institution - 0193, Jerusalem
  - Local Institution, Jerusalem
  - Local Institution - 0078, Jerusalem
  - Local Institution - 0308, Nahariya
  - Local Institution - 0247, Petah Tikva
  - Local Institution - 0204, Ramat Gan
  - Local Institution - 0086, Tel Aviv
- Italy (14):
  - Local Institution - 0359, Genoa, Liguria
  - Local Institution - 0084, Pavia, Lombardy
  - Local Institution - 0151, Ancona, The Marches
  - Local Institution - 0149, Negrar, Veneto
  - Local Institution - 0156, Bologna
  - Local Institution - 0290, Cagliari
  - Local Institution - 0095, Milan
  - Local Institution - 0104, Modena
  - Local Institution - 0085, Perugia
  - Local Institution - 0114, Perugia
  - Local Institution - 0108, Roma
  - Local Institution - 0129, Roma
  - Local Institution - 0083, Verona
  - Local Institution - 0123, Vibo Valentia
- Japan (53):
  - Local Institution - 0335, Kasugai, Aichi-ken
  - Local Institution - 0274, Nagoya, Aichi-ken
  - Local Institution - 0331, Toyoake Shi, Aichi-ken
  - Local Institution - 0325, Toyohashi, Aichi-ken
  - Local Institution - 0317, Toyota-shi, Aichi-ken
  - Local Institution - 0336, Sakura-shi, Chiba
  - Local Institution - 0320, Chikushino-shi, Fukuoka
  - Local Institution - 0259, Kasuga-shi, Fukuoka
  - Local Institution - 0311, Kitakyushu, Fukuoka
  - Local Institution - 0229, Kitakyushu-shi, Fukuoka
  - Local Institution - 0270, Kitakyushu-shi, Fukuoka
  - Local Institution - 0230, Koga-shi, Fukuoka
  - Local Institution - 0324, Kurume, Fukuoka
  - Local Institution - 0257, Aizuwakamatsu-shi, Fukushima
  - Local Institution - 0309, Takayama-shi, Gifu
  - Local Institution - 0211, Isesaki-shi, Gunma
  - Local Institution - 0337, Aki-gun, Hiroshima
  - Local Institution - 0240, Higashihiroshima-shi, Hiroshima
  - Local Institution - 0328, Hiroshima, Hiroshima
  - Local Institution - 0226, Kobe, Hyōgo
  - Local Institution - 0323, Kanazawa, Ishikawa-ken
  - Local Institution - 0446, Komatsu, Ishikawa-ken
  - Local Institution - 0299, Kagoshima, Kagoshima-ken
  - Local Institution - 0310, Kawasaki, Kanagawa
  - Local Institution - 0228, Kawasaki, Kanagawa
  - Local Institution - 0296, Sendai, Miyagi
  - Local Institution - 0278, Sendai, Miyagi
  - Local Institution - 0261, Nagasaki, Nagasaki
  - Local Institution - 0272, Izumisano, Osaka
  - Local Institution, Kishiwada, Osaka
  - Local Institution - 0279, Matsubara, Osaka
  - Local Institution - 0322, Sakai-shi, Osaka
  - Local Institution - 0251, Suita, Osaka
  - Local Institution - 0244, Suita-shi, Osaka
  - Local Institution - 0263, Hidaka, Saitama
  - Local Institution - 0334, Shimotsuke-shi, Tochigi
  - Local Institution - 0232, Bunkyo-ku, Tokyo
  - Local Institution - 0343, Hachiōji, Tokyo
  - Local Institution - 0255, Meguro-ku, Tokyo
  - Local Institution - 0338, Minato-ku, Tokyo
  - Local Institution - 0342, Minato-ku, Tokyo
  - Local Institution - 0295, Mitaka-shi, Tokyo
  - Local Institution - 0298, Shinagawa-ku, Tokyo
  - Local Institution - 0316, Shinjuku-ku, Tokyo
  - Local Institution - 0318, Tachikawa-shi, Tokyo
  - Local Institution - 0319, Shimonoseki-Shi, Yamaguchi
  - Local Institution - 0271, Fukuoka
  - Local Institution - 0243, Fukuoka
  - Local Institution - 0312, Kyoto
  - Local Institution - 0327, Osaka
  - Local Institution - 0239, Osaka
  - Local Institution - 0313, Osaka
  - Local Institution - 0301, Saga
- Mexico (6):
  - Local Institution - 0396, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution - 0398, Mexico City, Mexico City
  - Local Institution - 0404, Monterrey, Nuevo León
  - Local Institution - 0394, Culiacán, Sinaloa
  - Local Institution - 0366, Durango
- Norway (6):
  - Local Institution - 0368, Bergen
  - Local Institution - 0383, Grålum
  - Local Institution, Kristiansand
  - Local Institution - 0130, Lørenskog
  - Local Institution - 0408, Oslo
  - Local Institution - 0330, Stavanger
- Poland (15):
  - Local Institution - 0265, Warsaw, Masovian Voivodeship
  - Local Institution - 0350, Bydgoszcz
  - Local Institution - 0216, Chełm
  - Local Institution - 0206, Gdansk
  - Local Institution, Gmina Końskie
  - Local Institution - 0181, Grodzisk Mazowieciki
  - Local Institution - 0253, Katowice
  - Local Institution - 0197, Lodz
  - Local Institution - 0198, Olsztyn
  - Local Institution - 0215, Sandomierz
  - Local Institution - 0183, Skarżysko-Kamienna
  - Local Institution, Warsaw
  - Local Institution - 0214, Warsaw
  - Local Institution - 0225, Wałcz
  - Local Institution - 0212, Wejherowo
- Russia (8):
  - Local Institution - 0277, Barnaul
  - Local Institution - 0260, Kemerovo
  - Local Institution - 0306, Moscow
  - Local Institution, Moscow
  - Local Institution - 0268, Novosibirsk
  - Local Institution - 0356, Saint Petersburg
  - Local Institution - 0202, Smolensk
  - Local Institution, Yaroslavl
- South Korea (20):
  - Local Institution - 0094, Goyang-si, Gyeonggido
  - Local Institution - 0088, Seoul, Seoul Teugbyeolsi
  - Local Institution - 0081, Anyang
  - Local Institution - 0109, Busan
  - Local Institution - 0166, Busan
  - Local Institution - 0179, Daegu
  - Local Institution - 0102, Daegu
  - Local Institution, Daegu
  - Local Institution - 0105, Gwangju
  - Local Institution - 0101, Incheon
  - Local Institution - 0153, Seongnam-si
  - Local Institution - 0087, Seoul
  - Local Institution - 0185, Seoul
  - Local Institution - 0071, Seoul
  - Local Institution - 0080, Seoul
  - Local Institution - 0120, Seoul
  - Local Institution - 0145, Seoul
  - Local Institution - 0152, Seoul
  - Local Institution - 0112, Seoul
  - Local Institution - 0091, Seoul
- Spain (26):
  - Local Institution - 0159, Sabadell, Barcelona
  - Local Institution - 0163, Sant Joan Despí, Barcelona
  - Local Institution - 0372, León, Castille and León
  - Local Institution - 0141, A Coruña
  - Local Institution - 0026, Albacete
  - Local Institution - 0052, Badalona
  - Local Institution - 0012, Barcelona
  - Local Institution - 0010, Barcelona
  - Local Institution - 0027, Barcelona
  - Local Institution - 0385, Córdoba
  - Local Institution - 0400, Donostia / San Sebastian
  - Local Institution - 0426, Girona
  - Local Institution - 0176, L'Hospitalet de Llobregat
  - Local Institution - 0249, Lleida
  - Local Institution - 0238, Madrid
  - Local Institution - 0025, Madrid
  - Local Institution - 0413, Madrid
  - Local Institution - 0384, Madrid
  - Local Institution - 0425, Santiago de Compostela
  - Local Institution - 0158, Seville
  - Local Institution - 0177, Seville
  - Local Institution - 0164, Tarragona
  - Local Institution - 0150, Terrassa
  - Local Institution - 0147, Valencia
  - Local Institution - 0014, Valladolid
  - Local Institution - 0418, Vigo
- Sweden (5):
  - Local Institution - 0128, Malmo, Skåne County
  - Local Institution - 0171, Gothenburg
  - Local Institution - 0191, Hässleholm
  - Local Institution - 0224, Umeå
  - Local Institution - 0132, Uppsala
- Switzerland (6):
  - Local Institution - 0118, Basel, Basel-Stadt (de)
  - Local Institution - 0115, Bern, Bern (de)
  - Local Institution - 0162, Aarau
  - Local Institution - 0203, Geneva
  - Local Institution - 0201, Lausanne
  - Local Institution, Zurich
- United Kingdom (14):
  - Local Institution - 0222, Canterbury, Kent
  - Local Institution - 0140, Aberdeen
  - Local Institution, Ashford
  - Local Institution - 0157, Bath
  - Local Institution - 0089, Chester
  - Local Institution - 0221, Edinburgh
  - Local Institution - 0096, Glasgow
  - Local Institution - 0361, Lancashire
  - Local Institution, London
  - Local Institution - 0303, Luton
  - Local Institution, Nottingham
  - Local Institution - 0431, Salford
  - Local Institution - 0414, Sheffield
  - Local Institution - 0307, Staffordshire

REFERENCES:
- [Derived] Sharma M, Molina CA, Toyoda K, Bereczki D, Bangdiwala SI, Kasner SE, Lutsep HL, Tsivgoulis G, Ntaios G, Czlonkowska A, Shuaib A, Amarenco P, Endres M, Yoon BW, Tanne D, Toni D, Yperzeele L, von Weitzel-Mudersbach P, Sampaio Silva G, Avezum A, Dawson J, Strbian D, Tatlisumak T, Eckstein J, Ameriso SF, Weber JR, Sandset EC, Goar Pogosova N, Lavados PM, Arauz A, Gailani D, Diener HC, Bernstein RA, Cordonnier C, Kahl A, Abelian G, Donovan M, Pachai C, Li D, Hankey GJ. Safety and efficacy of factor XIa inhibition with milvexian for secondary stroke prevention (AXIOMATIC-SSP): a phase 2, international, randomised, double-blind, placebo-controlled, dose-finding trial. Lancet Neurol. 2024 Jan;23(1):46-59. doi: 10.1016/S1474-4422(23)00403-9. PMID 38101902
- [Derived] Whiteson HZ, Frishman WH. Factor XI/XIa Inhibitors: A New Approach to Anticoagulation. Cardiol Rev. 2025 Jul-Aug 01;33(4):306-311. doi: 10.1097/CRD.0000000000000624. Epub 2023 Dec 1. PMID 38038437
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Loading dose of Clopidogrel 300 mg + Aspirin 100 mg followed by Placebo + Aspirin 100 mg QD + Clopidogrel 75 mg QD on days 1-21 and Placebo + Aspirin 100 mg QD on days 22-90. All administered orally.
- Milvexian 25 mg QD: Loading dose of Clopidogrel 300 mg + Aspirin 100 mg followed by Milvexian 25 mg QD + Aspirin 100 mg QD + Clopidogrel 75 mg QD on days 1-21 and Milvexian 25 mg QD + Aspirin 100 mg QD on days 22-90. All administered orally.
- Milvexian 25 mg BID: Loading dose of Clopidogrel 300 mg + Aspirin 100 mg followed by Milvexian 25 mg BID + Aspirin 100 mg QD + Clopidogrel 75 mg QD on days 1-21 and Milvexian 25 mg BID + Aspirin 100 mg QD on days 22-90. All administered orally.
- Milvexian 50 mg BID: Loading dose of Clopidogrel 300 mg + Aspirin 100 mg followed by Milvexian 50 mg BID + Aspirin 100 mg QD + Clopidogrel 75 mg QD on days 1-21 and Milvexian 50 mg BID + Aspirin 100 mg QD on days 22-90. All administered orally.
- Milvexian 100 mg BID: Loading dose of Clopidogrel 300 mg + Aspirin 100 mg followed by Milvexian 100 mg BID + Aspirin 100 mg QD + Clopidogrel 75 mg QD on days 1-21 and Milvexian 100 mg BID + Aspirin 100 mg QD on days 22-90. All administered orally.
- Milvexian 200 mg BID: Loading dose of Clopidogrel 300 mg + Aspirin 100 mg followed by Milvexian 200 mg BID + Aspirin 100 mg QD + Clopidogrel 75 mg QD on days 1-21 and Milvexian 200 mg BID + Aspirin 100 mg QD on days 22-90. All administered orally.
- Milvexian 50 mg QD: Loading dose of Clopidogrel 300 mg + Aspirin 100 mg followed by Milvexian 50 mg QD + Aspirin 100 mg QD + Clopidogrel 75 mg QD on days 1-21 and Milvexian 50 mg QD + Aspirin 100 mg QD on days 22-90. All administered orally.
- Milvexian 100 mg QD: Loading dose of Clopidogrel 300 mg + Aspirin 100 mg followed by Milvexian 100 mg QD + Aspirin 100 mg QD + Clopidogrel 75 mg QD on days 1-21 and Milvexian 100 mg QD + Aspirin 100 mg QD on days 22-90. All administered orally.
Period: Randomization
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Started | 691 | 328 | 318 | 328 | 310 | 351 | 22 | 18
Completed | 682 | 324 | 313 | 325 | 306 | 345 | 22 | 17
Not Completed | 9 | 4 | 5 | 3 | 4 | 6 | 0 | 1
Not completed — Other reasons | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participant no longer meets study criteria | 5 | 3 | 4 | 0 | 2 | 3 | 0 | 1
Not completed — Participant request to discontinue study treatment | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Participant withdrew consent | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0
Period: Treatment
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Started | 682 | 325 (1 participant was randomized to Milvexian 200 mg BID, but received Milvexian 25 mg QD.) | 313 | 325 | 306 | 344 (1 participant was randomized to Milvexian 200 mg BID, but received Milvexian 25 mg QD.) | 22 | 17
Completed | 529 | 260 | 242 | 251 | 230 | 240 | 15 | 14
Not Completed | 153 | 65 | 71 | 74 | 76 | 104 | 7 | 3
Not completed — Adverse Event | 82 | 44 | 47 | 46 | 50 | 77 | 5 | 2
Not completed — Participant request to discontinue treatment | 34 | 6 | 10 | 10 | 14 | 15 | 0 | 1
Not completed — Participant withdrew consent | 11 | 4 | 5 | 5 | 4 | 4 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Poor/Non compliance | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Participant no longer meets study criteria | 9 | 1 | 5 | 4 | 4 | 4 | 2 | 0
Not completed — Other reasons | 13 | 8 | 3 | 7 | 3 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD | Total
Number analyzed (Participants) | 691 | 328 | 318 | 328 | 310 | 351 | 22 | 18 | 2366
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.1 (10.58) | 70.9 (10.66) | 70.1 (11.34) | 69.3 (10.69) | 69.7 (10.59) | 69.5 (11.11) | 65.7 (10.64) | 65.4 (11.65) | 69.6 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254 | 109 | 118 | 121 | 112 | 128 | 7 | 10 | 859
  Male | 437 | 219 | 200 | 207 | 198 | 223 | 15 | 8 | 1507
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 4 | 2 | 1 | 2 | 1 | 1 | 1 | 22
  Not Hispanic or Latino | 62 | 20 | 22 | 23 | 29 | 27 | 7 | 7 | 197
  Unknown or Not Reported | 619 | 304 | 294 | 304 | 279 | 323 | 14 | 10 | 2147
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 549 | 257 | 246 | 260 | 251 | 288 | 18 | 15 | 1884
    Black or African American | 15 | 5 | 6 | 8 | 3 | 5 | 3 | 3 | 48
    Asian | 35 | 12 | 21 | 13 | 11 | 17 | 0 | 0 | 109
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
    Asian Indian | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 6
    Chinese | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Japanese | 84 | 46 | 40 | 41 | 39 | 40 | 0 | 0 | 290
    Malay | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Asian Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Other | 5 | 6 | 2 | 4 | 5 | 1 | 1 | 0 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Model Based Assessment of Composite of New Ischemic Stroke During Treatment and New Covert Brain Infarction (FLAIR + DWI) Detected by MRI by Day 90
Description: Model based assessment estimate for composite event is a customized statistical analysis called MCP-MOD (Multiple Comparison Procedures, MODel) estimation, which is used to check for dose-response relationship. 95% confidence interval (CI) for composite event based on bootstrap (10000 samples).
Time Frame: From randomization to up to 90 days after randomization
Population: All randomized participants who experienced a new ischemic stroke by day 90, or an evaluable day 90 MRI regardless of when the MRI was collected. Dose -response model-based endpoint that was pre-specified for data to be collected only in the Placebo, 25 mg QD, and BID dose regimens.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID
Number analyzed (Participants) | 625 | 308 | 287 | 306 | 277 | 317
Percentage of participants | 16.8 [14.2 to 19.4] | 16.7 [14.4 to 19.0] | 16.6 [14.5 to 18.7] | 15.6 [13.6 to 17.9] | 15.4 [13.0 to 18.0] | 15.3 [12.3 to 20.4]
Statistical Analysis 1: Comparison: Placebo vs Milvexian 25 mg QD; Milvexian 25 mg QD over Placebo; Test type: Superiority; MCP-MOD; Multiple Comparison Procedures, MODel; Relative Risk (RR) = 0.99, 95% CI 2-sided [0.87 to 1.10] — 95% confidence interval (CI) for composite event based on bootstrap (10000 samples)
Statistical Analysis 2: Comparison: Placebo vs Milvexian 25 mg BID; Milvexian 25 mg BID over Placebo; Test type: Superiority; MCP-MOD; Multiple Comparison Procedures, MODel; Relative Risk (RR) = 0.99, 95% CI 2-sided [0.83 to 1.15] — 95% confidence interval (CI) for composite event based on bootstrap (10000 samples)
Statistical Analysis 3: Comparison: Placebo vs Milvexian 50 mg BID; Milvexian 50 mg BID over Placebo; Test type: Superiority; MCP-MOD; Multiple Comparison Procedures, MODel; Relative Risk (RR) = 0.93, 95% CI 2-sided [0.76 to 1.16] — 95% confidence interval (CI) for composite event based on bootstrap (10000 samples)
Statistical Analysis 4: Comparison: Placebo vs Milvexian 100 mg BID; Milvexian 100 mg BID over Placebo; Test type: Superiority; MCP-MOD; Multiple Comparison Procedures, MODel; Relative Risk (RR) = 0.92, 95% CI 2-sided [0.73 to 1.18] — 95% confidence interval (CI) for composite event based on bootstrap (10000 samples)
Statistical Analysis 5: Comparison: Placebo vs Milvexian 200 mg BID; Milvexian 200 mg BID over Placebo; Test type: Superiority; MCP-MOD; Multiple Comparison Procedures, MODel; Relative Risk (RR) = 0.91, 95% CI 2-sided [0.69 to 1.31] — 95% confidence interval (CI) for composite event based on bootstrap (10000 samples)

2. Secondary Outcome: Percent of Participants With Major Bleeding According to BARC Type 3 and 5
Description: Percent of participants with major bleeding based on the Bleeding Academic Research Consortium (BARC) Types 3 and 5 definitions. BARC bleeding types:
  3a = Overt bleeding plus hemoglobin drop of 3 to < 5 g/dL transfusion with overt bleeding 3b = Overt bleeding plus hemoglobin drop ≥5 g/dL; cardiac tamponade; bleeding requiring surgical intervention for control; bleeding requiring IV vasoactive agents 3c = Intracranial hemorrhage, 5a = Probable fatal bleeding 5b = Definite fatal bleeding
Time Frame: From first dose to up to 107 days after first dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 682 | 325 | 313 | 325 | 306 | 344 | 22 | 17
Percentage of participants | 0.6 [0.2 to 1.5] | 0.6 [0.1 to 2.2] | 0.6 [0.1 to 2.3] | 1.5 [0.5 to 3.6] | 1.6 [0.5 to 3.8] | 1.5 [0.5 to 3.4] | 0 [0 to 15.4] | 0 [0 to 19.5]

3. Secondary Outcome: Number of Participants With Bleeding Based on BARC Types 1-5
Description: Number of participants with bleeding based on Bleeding Academic Research Consortium (BARC) Type 1 to 5. BARC bleeding types: 0=No bleeding. 1=Not actionable bleeding. 2=Overt, actionable sign of hemorrhage requiring nonsurgical, medical intervention by a health-care professional, leading to hospitalization or increased level of care, or prompting evaluation. 3a=Overt bleeding plus hemoglobin drop of 3 to < 5 g/dL. 3b=Overt bleeding plus hemoglobin drop ≥5 g/dL; cardiac tamponade; bleeding requiring surgical intervention; bleeding requiring IV vasoactive agents. 3c=Intracranial hemorrhage; intraocular bleed compromising vision. 4=CABG-related bleeding, perioperative intracranial bleeding within 48 hours, reoperation after closure of sternotomy to control bleeding, transfusion of ≥5 U whole blood or packed red blood cells within a 48-hour period, chest tube output more than or equal to 2L within a 24-hour period. 5a=Probable fatal bleeding. 5b=Definite fatal bleeding.
Time Frame: From first dose to up to 107 days after first dose
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 682 | 325 | 313 | 325 | 306 | 344 | 22 | 17
Participants
  Type 1 | 41 | 26 | 16 | 28 | 25 | 22 | 5 | 2
  Type 2 | 9 | 7 | 9 | 7 | 10 | 8 | 1 | 1
  Type 3A | 2 | 1 | 1 | 1 | 2 | 3 | 0 | 0
  Type 3B | 0 | 1 | 1 | 1 | 3 | 1 | 0 | 0
  Type 3C | 2 | 0 | 0 | 3 | 0 | 1 | 0 | 0
  Type 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Type 5A | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Type 5B | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Bleeding Based on ISTH-Defined Criteria
Description: Number of participants with bleeding based on International Society on Thrombosis and Hemostasis (ISTH). ISTH Bleeding Types: 1) Fatal bleeding and/or 2) Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome and/or 3) Bleeding causing a fall in hemoglobin level of ≥2 g/dL, or leading to transfusion of ≥2 units of whole blood or red cells.
Time Frame: From first dose to up to 107 days after first dose
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 682 | 325 | 313 | 325 | 306 | 344 | 22 | 17
Participants
  Major | 4 | 2 | 2 | 5 | 6 | 5 | 0 | 0
  Clinically Relevant Non-Major (CRNM) | 7 | 8 | 9 | 7 | 8 | 8 | 1 | 1
  Major or CRNM | 11 | 10 | 11 | 12 | 14 | 13 | 1 | 1
  Minor Bleed | 43 | 25 | 16 | 28 | 26 | 22 | 5 | 2

5. Secondary Outcome: Number of Participants With Bleeding Based on PLATO-Defined Criteria
Description: Number of participants with bleeding based on Platelet Inhibition and Patient Outcomes (PLATO) defined criteria. PLATO bleeding definitions:
  1. Major Life-threatening: Fatal, Intracranial, Intrapericardial with cardiac tamponade, Resulting in hypovolemic shock or severe hypotension that requires pressors or surgery, Clinically overt or apparent bleeding associated with decrease in hemoglobin >5 g/dL, Requiring transfusion of ≥4 U whole blood or packed red blood cells (PRBCs)
  2. Other Major: Significantly disabling (eg, intraocular with permanent vision loss), Associated drop in hemoglobin of 3 to 5 g/dL, Requiring transfusion of 2 to 3 U whole blood or PRBCs
  3. Any Major: Any one of the above criteria
  4. Minor: Bleeding that does not meet criteria for PLATO Major bleeding, and requiring medical intervention
Time Frame: From first dose to up to 107 days after first dose
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 682 | 325 | 313 | 325 | 306 | 344 | 22 | 17
Participants
  MAJOR LIFE-THREATENING | 2 | 1 | 1 | 4 | 3 | 2 | 0 | 0
  OTHER MAJOR BLEEDING | 2 | 1 | 1 | 1 | 2 | 3 | 0 | 0
  ANY MAJOR | 4 | 2 | 2 | 5 | 5 | 5 | 0 | 0
  MINOR | 7 | 6 | 7 | 7 | 9 | 9 | 0 | 1
  MINIMAL | 43 | 27 | 18 | 28 | 26 | 21 | 6 | 2

6. Secondary Outcome: Percent of Participants With Descriptive Assessment of Composite of New Ischemic Stroke During Treatment and New Covert Brain Infarction (FLAIR + DWI) Detected by MRI by Day 90
Description: Descriptive Assessment of Composite of New Ischemic Stroke During Treatment and New Covert Brain Infarction (FLAIR + DWI) Detected by MRI by Day 90.
Time Frame: From randomization to up to 90 days after randomization
Population: All randomized participants who experienced a new ischemic stroke by day 90, or an evaluable day 90 MRI regardless of when the MRI was collected.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 625 | 308 | 287 | 306 | 277 | 317 | 21 | 16
Percentage of participants | 16.6 | 16.2 | 18.5 | 14.1 | 14.8 | 16.4 | 19.0 | 18.8

7. Secondary Outcome: Composite of Percent of Participants With New Ischemic Stroke, MI and All Cause Death
Description: Composite of percent of participants of new ischemic stroke, (Myocardial Infarction) MI and all cause death.
Time Frame: From randomization to up to 90 days after randomization
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 691 | 328 | 318 | 328 | 310 | 351 | 22 | 18
Percentage of participants | 6.1 [4.3 to 7.9] | 5.2 [2.8 to 7.6] | 4.7 [2.4 to 7.0] | 4.9 [2.5 to 7.2] | 5.2 [2.7 to 7.6] | 9.4 [6.3 to 12.5] | 18.2 [2.1 to 34.3] | 5.6 [0 to 16.1]

8. Secondary Outcome: National Institutes of Health Stroke Scale (NIHSS)
Description: The NIHSS is an 11-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. The score for each ability is a number between 0 and 4, 0 being normal functioning and 4 being completely impaired. The patient's NIHSS score is calculated by adding the number for each element of the scale; 42 is the highest score possible. In the NIHSS, the higher the score, the more impaired a stroke participant is.
Time Frame: At baseline, on Days 21 and 90, and at the time of a new stroke event
Population: All randomized participants with a complete NIHSS assessment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 684 | 324 | 311 | 326 | 305 | 348 | 22 | 17
Score on a scale
  Baseline | 1.6 (1.87) | 1.7 (1.68) | 1.6 (1.73) | 1.6 (1.79) | 1.8 (1.81) | 1.6 (1.79) | 1.1 (1.44) | 2.0 (1.70)
  Day 21: number analyzed (Participants) | 624 | 294 | 280 | 301 | 271 | 314 | 18 | 16
  Day 21 | 0.9 (2.11) | 0.8 (1.35) | 0.8 (1.43) | 0.8 (1.58) | 0.8 (1.48) | 0.9 (1.88) | 0.8 (1.90) | 0.9 (1.39)
  Day 90: number analyzed (Participants) | 552 | 263 | 251 | 259 | 238 | 256 | 20 | 14
  Day 90 | 0.5 (1.40) | 0.6 (1.06) | 0.6 (1.51) | 0.6 (1.14) | 0.6 (1.32) | 0.6 (1.29) | 0.3 (0.72) | 0.6 (1.45)
  First recurrent stroke: number analyzed (Participants) | 29 | 14 | 11 | 11 | 10 | 20 | 3 | 1
  First recurrent stroke | 6.2 (5.01) | 4.6 (6.79) | 5.4 (3.17) | 4.6 (4.30) | 7.1 (4.68) | 4.4 (4.60) | 5.3 (3.06) | 1.0 (NA) — Insufficient number of participants with events

9. Secondary Outcome: Modified Rankin Scale (mRS)
Description: The Modified Rankin Score (mRS) is a 6-point disability scale with possible scores ranging from 0 to 6.
  0 = No symptoms at all
  1. = No significant disability despite symptoms; able to carry out all usual duties and activities
  2. = Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. = Moderate disability; requiring some help, but able to walk without assistance
  4. = Moderately severe disability; unable to walk and attend to bodily needs without assistance
  5. = Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. = Dead
Time Frame: At baseline, on Days 21 and 90, and at the time of a new stroke event
Population: All randomized participants with a complete mRS assessment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 688 | 326 | 314 | 328 | 309 | 349 | 22 | 17
Score on a scale
  Baseline | 0.5 (0.87) | 0.6 (0.95) | 0.6 (0.96) | 0.5 (0.86) | 0.5 (0.89) | 0.6 (0.95) | 0.2 (0.53) | 0.7 (0.99)
  Day 21: number analyzed (Participants) | 630 | 301 | 287 | 306 | 279 | 316 | 17 | 16
  Day 21 | 1.0 (1.18) | 1.0 (1.13) | 0.9 (1.15) | 0.9 (1.15) | 1.0 (1.17) | 0.9 (1.19) | 0.9 (1.27) | 1.3 (1.14)
  Day 90: number analyzed (Participants) | 562 | 269 | 257 | 265 | 245 | 259 | 20 | 14
  Day 90 | 0.7 (1.04) | 0.8 (1.04) | 0.8 (1.07) | 0.7 (1.01) | 0.7 (1.01) | 0.8 (1.05) | 0.6 (1.05) | 1.0 (1.11)
  First recurrent stroke: number analyzed (Participants) | 26 | 13 | 10 | 11 | 8 | 19 | 2 | 1
  First recurrent stroke | 3.0 (1.60) | 2.7 (1.03) | 2.6 (1.35) | 2.3 (1.62) | 2.9 (1.64) | 1.8 (1.72) | 2.0 (0.00) | 1.0 (NA) — Insufficient number of participants with events

10. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: The Montreal Cognitive Assessment (MoCA) is a survey with a summed score. MoCA score ranges between a lowest score of 0 to a highest score of 30. A score of:
  * ≥26 points: indicates normal cognitive function
  * 18-25 points: Mild cognitive impairment
  * 10-17 points: Moderate cognitive impairment
  * fewer than 10 points: Severe cognitive impairment
Time Frame: At baseline, on Days 21 and 90, and at the time of a new stroke event
Population: All randomized participants with a complete MoCA assessment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 541 | 257 | 235 | 257 | 235 | 276 | 17 | 14
Score on a scale
  Baseline | 22.3 (5.06) | 21.6 (5.59) | 22.0 (5.18) | 22.5 (4.82) | 22.4 (5.04) | 22.1 (5.31) | 24.4 (3.84) | 22.0 (4.59)
  Day 21: number analyzed (Participants) | 492 | 231 | 206 | 236 | 211 | 251 | 15 | 13
  Day 21 | 24.0 (4.77) | 23.9 (5.01) | 24.0 (4.70) | 24.3 (4.57) | 23.6 (4.48) | 24.0 (4.96) | 26.4 (2.61) | 24.1 (4.70)
  Day 90: number analyzed (Participants) | 435 | 208 | 183 | 209 | 180 | 210 | 15 | 11
  Day 90 | 24.6 (4.54) | 24.0 (4.69) | 24.2 (4.80) | 24.4 (4.48) | 24.5 (4.36) | 24.2 (5.05) | 25.0 (4.72) | 26.4 (1.69)
  First recurrent stroke: number analyzed (Participants) | 10 | 3 | 3 | 2 | 1 | 8 | 1 | 1
  First recurrent stroke | 23.2 (6.63) | 17.3 (6.11) | 25.3 (2.31) | 19.0 (8.49) | 3.0 (NA) — Insufficient number of participants with events | 23.1 (7.08) | 11.0 (NA) — Insufficient number of participants with events | 22.0 (NA) — Insufficient number of participants with events

11. Secondary Outcome: Digit Symbol Substitution Test (DSST)
Description: The Descriptive Summary of the Digit Symbol Substitution Test (DSST) is a scale item, with a lowest score of 0 and highest total score of 135. Higher score indicates better cognitive functioning.
Time Frame: At baseline, on Days 21 and 90, and at the time of a new stroke event
Population: All randomized participants with a complete DSST assessment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 493 | 238 | 209 | 234 | 220 | 257 | 17 | 14
Score on a scale
  Baseline | 34.9 (22.36) | 31.2 (18.87) | 32.9 (22.89) | 37.2 (25.67) | 33.7 (21.89) | 31.7 (19.15) | 47.1 (29.34) | 29.2 (18.16)
  Day 21: number analyzed (Participants) | 443 | 213 | 183 | 213 | 194 | 228 | 14 | 13
  Day 21 | 41.2 (22.14) | 38.9 (19.27) | 40.2 (21.60) | 45.1 (25.77) | 41.2 (22.87) | 39.1 (21.35) | 54.6 (32.73) | 37.1 (20.13)
  Day 90: number analyzed (Participants) | 394 | 191 | 160 | 186 | 166 | 192 | 15 | 11
  Day 90 | 42.8 (21.18) | 41.7 (21.66) | 41.3 (20.29) | 45.2 (21.86) | 45.5 (23.44) | 41.4 (21.97) | 47.5 (27.48) | 40.7 (17.46)
  First recurrent stroke: number analyzed (Participants) | 8 | 3 | 3 | 2 | 1 | 6 | 1 | 1
  First recurrent stroke | 36.3 (13.56) | 28.0 (20.95) | 42.0 (4.36) | 40.5 (2.12) | 23.0 (NA) — Insufficient number of participants with events | 27.5 (16.96) | 9.0 (NA) — Insufficient number of participants with events | 47.0 (NA) — Insufficient number of participants with events

12. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AE: include all non-serious adverse events with onset on or after first dose date and within 2 days after the last dose of study treatment.
Time Frame: From first dose to 2 days after last dose of study therapy (up to approximately 107 days)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 682 | 325 | 313 | 325 | 306 | 344 | 22 | 17
Participants | 399 | 190 | 186 | 192 | 193 | 211 | 11 | 13

13. Secondary Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities
Description: Number of participants with clinically significant vital sign abnormalities. Vital signs included heart rate and diastolic and systolic blood pressure.
Time Frame: From first dose to up to 90 days after first dose
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 682 | 325 | 313 | 325 | 306 | 344 | 22 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Abnormalities
Description: Number of participants with clinically significant physical examination abnormalities.
Time Frame: From first dose to up to 90 days after first dose
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 682 | 325 | 313 | 325 | 306 | 344 | 22 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Number of participants with clinically significant ECG abnormalities.
Time Frame: From first dose to up to 90 days after first dose
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 682 | 325 | 313 | 325 | 306 | 344 | 22 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities - Liver
Description: The number of treated participants who experienced a laboratory abnormality of the liver during the course of the study.
  Aspartate aminotransferase (AST) Alanine aminotransferase (ALT) Upper Limit of Normal (ULN) Results reported in International System of Units (SI)
Time Frame: From first dose to up to approximately 38 months
Population: All treated participants with at least one clinically significant liver laboratory abnormality
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 642 | 303 | 280 | 306 | 281 | 324 | 21 | 16
Participants
  ALT > 3x ULN: number analyzed (Participants) | 642 | 303 | 280 | 306 | 280 | 324 | 20 | 16
  ALT > 3x ULN | 4 | 2 | 0 | 2 | 3 | 3 | 0 | 0
  ALT > 5x ULN: number analyzed (Participants) | 642 | 303 | 280 | 306 | 280 | 324 | 20 | 16
  ALT > 5x ULN | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0
  ALT > 10x ULN: number analyzed (Participants) | 642 | 303 | 280 | 306 | 280 | 324 | 20 | 16
  ALT > 10x ULN | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  ALT > 20x ULN: number analyzed (Participants) | 642 | 303 | 280 | 306 | 280 | 324 | 20 | 16
  ALT > 20x ULN | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  AST > 3x ULN: number analyzed (Participants) | 641 | 302 | 280 | 304 | 281 | 323 | 21 | 16
  AST > 3x ULN | 6 | 5 | 1 | 4 | 3 | 3 | 1 | 0
  AST > 5x ULN: number analyzed (Participants) | 641 | 302 | 280 | 304 | 281 | 323 | 21 | 16
  AST > 5x ULN | 3 | 2 | 1 | 0 | 2 | 1 | 1 | 0
  AST > 10x ULN: number analyzed (Participants) | 641 | 302 | 280 | 304 | 281 | 323 | 21 | 16
  AST > 10x ULN | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  AST > 20x ULN: number analyzed (Participants) | 641 | 302 | 280 | 304 | 281 | 323 | 21 | 16
  AST > 20x ULN | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALP > 2x ULN: number analyzed (Participants) | 640 | 300 | 276 | 305 | 279 | 319 | 20 | 16
  ALP > 2x ULN | 4 | 5 | 1 | 6 | 4 | 2 | 0 | 0
  Total Bilirubin > 1.5x ULN: number analyzed (Participants) | 639 | 302 | 277 | 304 | 279 | 318 | 20 | 16
  Total Bilirubin > 1.5x ULN | 10 | 6 | 2 | 7 | 5 | 2 | 0 | 0
  Total Bilirubin > 2x ULN: number analyzed (Participants) | 639 | 302 | 277 | 304 | 279 | 318 | 20 | 16
  Total Bilirubin > 2x ULN | 3 | 1 | 1 | 2 | 2 | 1 | 0 | 0
  Concurrent ALT/AST Elevation > 3x ULN with total bilirubin >2x ULN: number analyzed (Participants) | 639 | 302 | 277 | 304 | 279 | 318 | 20 | 16
  Concurrent ALT/AST Elevation > 3x ULN with total bilirubin >2x ULN | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

17. Secondary Outcome: Percent Change From Baseline in aPTT Activity
Description: Percent change from baseline in activated partial thromboplastin time (aPTT) activity via exposure response.
Time Frame: Baseline and day 90
Population: All participants with at least one aPTT pharmacodynamic endpoint assessed after first dose
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 503 | 251 | 226 | 241 | 214 | 232 | 14 | 14
Percent change | 2.47 (0.768) | 38.72 (2.264) | 58.30 (3.195) | 97.32 (3.601) | 140.76 (5.154) | 193.64 (7.041) | 48.48 (11.243) | 118.06 (13.840)

18. Secondary Outcome: Percent Change From Baseline in Factor XI Clotting Activity
Description: Percent change from baseline in factor XI clotting activity via exposure response.
Time Frame: Baseline and day 90
Population: All participants with at least one factor XI clotting pharmacodynamic endpoint assessed after first dose
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 503 | 251 | 223 | 228 | 216 | 236 | 15 | 13
Percent change | 4.48 (3.455) | -8.88 (1.280) | -17.67 (1.900) | -37.20 (1.655) | -61.52 (1.869) | -70.25 (3.043) | 3.86 (13.754) | -44.27 (6.501)

19. Secondary Outcome: Pharmacokinetic Parameter - Estimated Clearance (CL)
Description: Pharmacokinetic Parameter - Estimated Clearance (CL). CL is derived from plasma concentration versus time data. PK parameters were generated using a Population Pharmacokinetics (PPK) model. Summary statistics for these individual predicted PK parameters and exposures were stratified by dose. The PPK model analysis was based on combined PK data collected on days 1, 21, and 90.
Time Frame: From first dose to up to 90 days after first dose
Population: All treated participants with at least one post-dose PK sample. Pre-specified for data to be collected only in the 25 mg QD, and BID dose regimens.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID
Number analyzed (Participants) | 323 | 307 | 323 | 303 | 341
L/h | 8.15 (34) | 8.01 (34.3) | 7.54 (32.8) | 7.08 (31.3) | 7.43 (32.9)

20. Secondary Outcome: Pharmacokinetic Parameter - Volume of the Central Compartment (VC)
Description: Pharmacokinetic Parameter - Volume of the Central Compartment (VC). VC is derived from plasma concentration versus time data. PK parameters were generated using a Population Pharmacokinetics (PPK) model. Summary statistics for these individual predicted PK parameters and exposures were stratified by dose. The PPK model analysis was based on combined PK data collected on days 1, 21, and 90.
Time Frame: From first dose to up to 90 days after first dose
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID
Number analyzed (Participants) | 323 | 307 | 323 | 303 | 341
L | 34.9 (152) | 31.4 (138) | 30.9 (145) | 28.9 (149) | 31.6 (181)

21. Secondary Outcome: Volume of Incident Infarcts (New DWI+ or DWI- Lesions) by Participant on Day 90 MRI
Description: Total volume of diffusion-weighted imaging (DWI) magnetic resonance imaging (MRI) infarcts on the DWI Sequence on day 90 MRI.
Time Frame: At day 90
Population: All randomized participants with an evaluable MRI
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 82 | 40 | 49 | 36 | 35 | 35 | 3 | 3
mL | 2.3492 (11.40906) | 0.8976 (1.96342) | 2.9902 (8.28993) | 1.2682 (2.72452) | 1.4727 (3.78795) | 1.2711 (4.05035) | 8.8960 (13.85294) | 1.4503 (1.89112)

22. Secondary Outcome: Number of Incident Infarcts (New DWI+ or DWI- Lesions) by Participant on Day 90 MRI
Description: Number of diffusion-weighted imaging (DWI) magnetic resonance imaging (MRI) infarcts on the DWI Sequence on day 90 MRI.
Time Frame: At day 90
Population: All randomized participants with an evaluable MRI
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 82 | 40 | 49 | 36 | 35 | 35 | 3 | 3
Participants
  >0 | 82 | 40 | 49 | 36 | 35 | 35 | 3 | 3
  1 | 57 | 26 | 36 | 26 | 24 | 23 | 1 | 2
  2 | 11 | 8 | 5 | 5 | 3 | 6 | 2 | 0
  3 | 8 | 5 | 4 | 1 | 2 | 2 | 0 | 0
  4 | 1 | 1 | 2 | 3 | 2 | 2 | 0 | 1
  5 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  >5 | 4 | 0 | 2 | 1 | 3 | 0 | 0 | 0

23. Other Pre Specified Outcome: Percent of Participants With Ischemic Stroke Events
Description: Secondary analysis of symptomatic ischemic stroke events. Clinical events are included up to day 90. Wald 95% CI within group. Undetermined stroke is included.
Time Frame: From randomization to up to 90 days after randomization
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID | Milvexian 50 mg QD | Milvexian 100 mg QD
Number analyzed (Participants) | 691 | 328 | 318 | 328 | 310 | 351 | 22 | 18
Percentage of participants
  Ischemic stroke | 5.5 [3.8 to 7.2] | 4.6 [2.3 to 6.8] | 3.8 [1.7 to 5.9] | 4.0 [1.9 to 6.1] | 3.5 [1.5 to 5.6] | 7.7 [4.9 to 10.5] | 13.6 [0.0 to 28.0] | 5.6 [0.0 to 16.1]
  Undetermined stroke | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Placebo vs Milvexian 25 mg QD; Milvexian 25 mg QD over Placebo; Test type: Superiority; Wald Confidence Limits; 95% CIs for RR are constructed using Wald Confidence Limits; Relative Risk (RR) = 0.83, 95% CI 2-sided [0.46 to 1.49]
Statistical Analysis 2: Comparison: Placebo vs Milvexian 25 mg BID; Milvexian 25 mg BID over Placebo; Test type: Superiority; Wald Confidence Limits; 95% CIs for RR are constructed using Wald Confidence Limits; Relative Risk (RR) = 0.69, 95% CI 2-sided [0.36 to 1.30]
Statistical Analysis 3: Comparison: Placebo vs Milvexian 50 mg BID; Milvexian 50 mg BID over Placebo; Test type: Superiority; Wald Confidence Limits; 95% CIs for RR are constructed using Wald Confidence Limits; Relative Risk (RR) = 0.72, 95% CI 2-sided [0.39 to 1.33]
Statistical Analysis 4: Comparison: Placebo vs Milvexian 100 mg BID; Milvexian 100 mg BID over Placebo; Test type: Superiority; Wald Confidence Limits; 95% CIs for RR are constructed using Wald Confidence Limits; Relative Risk (RR) = 0.65, 95% CI 2-sided [0.33 to 1.25]
Statistical Analysis 5: Comparison: Placebo vs Milvexian 200 mg BID; Milvexian 200 mg BID; Test type: Superiority; Wald Confidence Limits; 95% CIs for RR are constructed using Wald Confidence Limits; Relative Risk (RR) = 1.40, 95% CI 2-sided [0.87 to 2.25]
Statistical Analysis 6: Comparison: Placebo vs Milvexian 50 mg QD; Milvexian 50 mg QD over Placebo; Test type: Superiority; Wald Confidence Limits; 95% CIs for RR are constructed using Wald Confidence Limits; Relative Risk (RR) = 2.48, 95% CI 2-sided [0.83 to 7.42]
Statistical Analysis 7: Comparison: Placebo vs Milvexian 100 mg QD; Milvexian 100 mg QD over Placebo; Test type: Superiority; Wald Confidence Limits; 95% CIs for RR are constructed using Wald Confidence Limits; Relative Risk (RR) = 1.01, 95% CI 2-sided [0.15 to 6.96]

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their randomization until their study completion (up to approximately 38 months). SAEs and Other AEs were assessed from first dose to 7 days after last dose of study therapy (up to approximately 112 days).
Description: The total number at risk for all-cause mortality represents all participants who were randomized. The total number at risk by any serious adverse event and other (not including serious) adverse events represents all participants who received at least 1 dose of study medication.
Arm/Group | Placebo | Milvexian 25 mg QD | Milvexian 50 mg QD | Milvexian 100 mg QD | Milvexian 25 mg BID | Milvexian 50 mg BID | Milvexian 100 mg BID | Milvexian 200 mg BID
All-Cause Mortality (participants affected / at risk) | 5/691 | 4/328 | 0/22 | 0/18 | 3/318 | 3/328 | 5/310 | 5/351
Serious Adverse Events (participants affected / at risk) | 94/682 | 37/325 | 5/22 | 3/17 | 39/313 | 41/325 | 42/306 | 54/344
Other Adverse Events (participants affected / at risk) | 178/682 | 81/325 | 6/22 | 11/17 | 83/313 | 92/325 | 82/306 | 90/344
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=682) | Milvexian 25 mg QD (N=325) | Milvexian 50 mg QD (N=22) | Milvexian 100 mg QD (N=17) | Milvexian 25 mg BID (N=313) | Milvexian 50 mg BID (N=325) | Milvexian 100 mg BID (N=306) | Milvexian 200 mg BID (N=344)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 3 | 0 | 0 | 1 | 0 | 3 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nodal rhythm (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis fulminant (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 5 | 2 | 0 | 0 | 2 | 1 | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis intestinal perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infected dermal cyst (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0 | 1 | 0 | 0 | 1 | 2 | 1
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 5
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection pseudomonas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Reactive gastropathy (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basilar artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basilar artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basilar migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brain stem stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Carotid artery thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 4 | 1 | 0 | 0 | 1 | 0 | 1 | 2
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral venous thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Focal dyscognitive seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 3 | 1 | 0 | 0 | 3 | 2 | 1 | 3
Ischaemic stroke (Nervous system disorders) | 21 | 9 | 3 | 1 | 6 | 10 | 7 | 11
Lacunar stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myasthenia gravis crisis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudostroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sedation complication (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Stroke in evolution (Nervous system disorders) | 5 | 2 | 0 | 1 | 4 | 1 | 1 | 8
Syncope (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 8 | 1 | 0 | 0 | 4 | 1 | 4 | 4
Vertebral artery dissection (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Malignant hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=682) | Milvexian 25 mg QD (N=325) | Milvexian 50 mg QD (N=22) | Milvexian 100 mg QD (N=17) | Milvexian 25 mg BID (N=313) | Milvexian 50 mg BID (N=325) | Milvexian 100 mg BID (N=306) | Milvexian 200 mg BID (N=344)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 0 | 2 | 2 | 2 | 5 | 8
Increased tendency to bruise (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 3 | 0 | 1 | 0 | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 44 | 22 | 0 | 3 | 17 | 20 | 20 | 24
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 14 | 11 | 1 | 2 | 6 | 6 | 11 | 5
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 7 | 7 | 0 | 1 | 2 | 3 | 3 | 3
Fatigue (General disorders) | 6 | 2 | 0 | 2 | 3 | 1 | 2 | 4
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 0
Thirst (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 17 | 8 | 0 | 1 | 9 | 6 | 11 | 12
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1 | 3 | 1 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1 | 0 | 2 | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 7 | 4 | 0 | 1 | 4 | 7 | 5 | 2
Headache (Nervous system disorders) | 23 | 16 | 3 | 1 | 12 | 14 | 12 | 9
Paraesthesia (Nervous system disorders) | 3 | 0 | 1 | 2 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 0
Tremor (Nervous system disorders) | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 5 | 3 | 1 | 1 | 6 | 3 | 5 | 3
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0 | 2 | 1 | 1 | 1 | 9
Pollakiuria (Renal and urinary disorders) | 2 | 1 | 0 | 1 | 0 | 1 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 2 | 0 | 4 | 5 | 4 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 56 | 21 | 0 | 2 | 23 | 24 | 20 | 19
Hypotension (Vascular disorders) | 5 | 2 | 0 | 1 | 2 | 4 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT03766581/Prot_SAP_000.pdf